CLINICAL TRIAL: NCT05828719
Title: Randomized Controlled Trial of Revascularization Versus Medical Treatment on Clinical Outcomes in Patients With Reduced Left Ventricular Function
Brief Title: Revascularization Versus Medical Treatment in Patients With Ischemic Left Ventricular Dysfunction
Acronym: RESTORE-PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Bin Song, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESTORE119023
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Ischemic Cardiomyopathy
Keywords: ischemic cardiomyopathy; percutaneous coronary intervention; ejection fraction; guideline-directed medical treatment
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label, randomized controlled, superiority trial
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guideline-directed medical treatment group (No Intervention): In the GDMT group, medical treatment for patients with left ventricular dysfunction will be performed under current ACC/AHA/SCAI or ESC/EACTS guidelines for heart failure.
- Revascularization group (Experimental): In the revascularization group, patients will undergo percutaneous coronary intervention (PCI) using standard techniques under current ACC/AHA/SCAI or ESC/EACTS guidelines. In the revascularization group, the procedure must be within 2 weeks of randomization.
  Revascularization criteria is presented as below. Revascularization indication
  1. Diameter stenosis >90% by visual assessment
  2. Functionally significant stenosis (FFR≤0.80 or non-hyperemic pressure ratios≤0.89)
  3. Chronic total occlusion with substantial ischemic territory. The below locations will be judged as having substantial ischemic territory.
     * Left main artery
     * Proximal to mid left anterior descending artery
     * Proximal left circumflex artery in left dominant coronary arterial system
     * Proximal to distal right coronary artery in right dominant coronary arterial system
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Revascularization indication
  1. Diameter stenosis >90% by visual assessment
  2. Functionally significant stenosis (FFR≤0.80 or non-hyperemic pressure ratios≤0.89)
  3. Chronic total occlusion with substantial ischemic territory. The below locations will be judged as having substantial ischemic territory.
     * Left main artery
     * Proximal to mid left anterior descending artery
     * Proximal left circumflex artery in left dominant coronary arterial system
     * Proximal to distal right coronary artery in right dominant coronary arterial system
  Arms: Revascularization group

SUMMARY:
Randomized trial to compare clinical outcomes between revascularization versus medical treatment alone in patients with ischemic cardiomyopathy and left ventricular dysfunction.

DETAILED DESCRIPTION:
Ischemic cardiomyopathy, the term used to describe systolic dysfunction due to chronic myocardial ischemia from ischemic heart disease, is the most common form of heart failure. To adapt to this ischemic environment, myocardium is known to undergo downregulation that may revert after adequate perfusion is re-established, a phenomenon known as myocardium hibernation. This phenomenon has been a background for the main concept of management for ischemic cardiomyopathy via revascularization. Indeed, the recent 10-year follow-up reports from STICH trial demonstrated improved long-term clinical outcomes after coronary bypass graft surgery than optimal medical therapy (OMT) in patients with ischemic cardiomyopathy.

Percutaneous coronary intervention (PCI) is another intervention that is commonly used to revascularize significant coronary stenosis. Despite common belief that revascularization by PCI would improve perfusion to ischemic myocardium and improve clinical outcomes, several clinical trials have failed to show beneficial impact of PCI over OMT in stable ischemic heart disease other than symptomatic improvement. Recently published REVIVED trial compared effect of PCI and OMT in ischemic cardiomyopathy patients with left ventricular ejection fraction < 35% and demonstrable viable myocardial segments, and found no significant difference in clinical outcomes of both groups.

However, whether PCI optimized by additional information can make a difference in this setting remains unanswered. It is known that intravascular imaging and coronary physiologic testing using intravascular ultrasound (IVUS), optical coherence tomography (OCT) or fractional flow reserve (FFR) result in better outcomes compared to conventional angiography alone. IVUS provides anatomical information regarding the lumen, plaque, and plaque characteristics, and can optimize stent placement minimizing stent-related problems and lead to better outcomes. On the other hand, FFR provides information on amount of ischemia which the stenosis in question is causing, and also improves the quality of PCI which has been demonstrated by multiple previous trials. Unfortunately, proportion of IVUS and FFR use is not disclosed in REVIVED trial, and it is possible there is a room for improvement if the PCI is further guided by these adjunctive diagnostic procedures in regard to the clinical outcomes.

In this regard, it is our hypothesis that PCI guided and optimized by intravascular imaging and FFR-guided strategy would bring additional benefit that may result in significant difference of prognosis for ischemic cardiomyopathy compared to OMT alone. Randomized controlled trial to test this hypothesis would provide valuable evidence to guide treatment strategy for ischemic cardiomyopathy. Therefore, RESTORE-PCI trial has been designed to compare clinical outcomes after state-of-the-art PCI or OMT for ischemic cardiomyopathy.

The aim of the study is to compare clinical outcomes between revascularization versus medical treatment alone in patients with ischemic cardiomyopathy and left ventricular dysfunction. Primary hypothesis is that revascularization guided by invasive physiologic indexes and optimized by intravascular imaging device plus optimal medical treatment (OMT) would reduce risk of primary composite end point (major adverse cardiac events [MACE], a composite of death, myocardial infarction (MI), admission for heart failure, or advanced heart failure requiring LVAD or transplantation) than OMT alone in patients with ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age
* Patients with stage C heart failure and left ventricular ejection fraction<40%
* Patients with significant coronary artery stenosis (diameter stenosis>50% with proven inducible myocardial ischemia by invasive physiologic assessment)
* Coronary artery disease is amenable for percutaneous coronary intervention (PCI)
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive approach and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Myocardial infarction by universal definition within 4 weeks of randomization
* Non-viable myocardium in myocardial viability test (cardiac magnetic resonance, dobutamine-stress echocardiography, delayed single-photon emission computerized tomography, or aneurysmal change in echocardiography)
* Target lesions not amenable for PCI by operators' decision
* Patients who need left ventricular assisted device (LVAD) or heart transplantation at the time of randomization
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, or Everolimus
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Pregnancy or breast feeding
* Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac events [MACE] | 2 years after last patient enrollment
  a composite of death, myocardial infarction (MI), admission for heart failure, or advanced heart failure requiring LVAD or transplantation

SECONDARY OUTCOMES:
All-cause death | 2 years after last patient enrollment
  All-cause death
Cardiac death | 2 years after last patient enrollment
  Cardiac death
Any myocardial infarction | 2 years after last patient enrollment
  Any myocardial infarction by Forth Universal definition of MI
Spontaneous myocardial infarction | 2 years after last patient enrollment
  Spontaneous myocardial infarction by Forth Universal definition of MI
Procedure-related myocardial infarction | After index procedure
  Procedure-related myocardial infarction by ARC II definition
Admission for heart failure | 2 years after last patient enrollment
  Admission for acute decompensated heart failure
Advanced heart failure requiring LVAD or transplantation | 2 years after last patient enrollment
  Advanced heart failure requiring LVAD or transplantation
Implantable cardioverter-defibrillator (ICD) or Cardiac resynchronization therapy (CRT-D) | 2 years after last patient enrollment
  Incidence of Implantable cardioverter-defibrillator (ICD) or Cardiac resynchronization therapy (CRT-D) for documented ventricular tachycardia or ventricular fibrillation (secondary prevention).
Clinically-indicated unplanned revascularization | 2 years after last patient enrollment
  Clinically-indicated unplanned revascularization
Stroke | 2 years after last patient enrollment
  Stroke (ischemic or hemorrhagic)
EQ-5D-5L (quality of life) | at 6 month after index procedure
  EQ-5D-5L (quality of life)
SAQ (angina severity) | at 6 month after index procedure
  SAQ (angina severity)
Left ventricular ejection fraction | at 6 month - 1 year follow-up after index procedure
  Left ventricular ejection fraction by echocardiography
NT-proBNP | at 6 month - 1 year follow-up after index procedure
  NT-proBNP, pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Young Bin Song, MD, PhD, Study Chair — Samsung Medical Center; Young Bin Song, MD, PhD, Principal Investigator — Samsung Medical Center; Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsune Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, SAP
Time Frame: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked